CLINICAL TRIAL: NCT04197349
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Phase 1 Study to Determine the Safety, Tolerability, and Pharmacokinetics of ALD1910, a Humanized Anti-Pituitary Adenylate Cyclase Activating Peptide (PACAP) Monoclonal Antibody
Brief Title: Safety, Tolerability and Pharmacokinetics of ALD1910 in Healthy Men and Woman
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Alder Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ALD1910-CLIN-001; 18902A (Other: H. Lundbeck A/S)
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A Cohort 1-8 (Experimental): ALD1910/Placebo; Single Dose IV infusion on Day 1
  Interventions: Biological: ALD1910
- Part B Cohort 9 (Experimental): ALD1910/Placebo+Sumatriptan; Single Dose IV infusion on Day 1
  Interventions: Biological: ALD1910; Biological: Sumatriptan
- Part B Cohort 10 (Experimental): ALD1910/Placebo; Single dose subcutaneous injection on Day 1
  Interventions: Biological: ALD1910

INTERVENTIONS:
Biological: ALD1910 — Single Dose IV infusion
  Arms: Part A Cohort 1-8; Part B Cohort 9
Biological: Sumatriptan — Single dose subcutaneous injection
  Arms: Part B Cohort 9
Biological: ALD1910 — Single dose subcutaneous injection
  Arms: Part B Cohort 10

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics of ALD1910, a monoclonal antibody, administered by intravenous infusion and subcutaneous injection.

DETAILED DESCRIPTION:
This is a first-in-humam, randomized, double-blind, placebo-controlled study in a healthy population. Up to 7 single ascending doses (cohorts 1 to 7) will be studied to determine the safety and tolerability of ALD1910. Approximately 96 healthy male and female participants are planned for the study, 64 for Part A and 32 for Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female
2. All female subjects must have a negative pregnancy test result and subjects to use of adequate contraception for the duration of the study.
3. Body Mass Index (BMI) between 18.0 and 30.0 kg/m2, and a total body weight of 50 to 100 kg inclusive.

Exclusion Criteria:

1. Use of prescription meds, nutritional supplements, OTC medications.
2. New or unusually strenuous exercise for the duration of the trial.
3. Current or previous drug or alcohol abuse.
4. Current, or previous smoker within 12 weeks prior to screening. Causal or social smokers are allowed.
5. Previous treatment or clinical trial with a monoclonal antibody 6 months prior to screening.
6. Current participation in any clinical research study.
7. ECG QTcF greater than or equal to 450 msec.
8. Greater than 6.4% glycosylated hemoglobin (HgbA1c) at screening
9. Fasting blood glucose greater than or equal to 126 mg/dL (7 mmol/L) at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events | From dosing to week 20
  Safety and tolerability based on the safety assessments (clinical safety laboratory tests, vital signs, ECG parameters)

SECONDARY OUTCOMES:
Area under the serum concentration-time curve (AUC(0-T)) | From dosing to week 20
Peak serum concentration (Cmax) | From dosing to week 20
Clearance (Cl) | From dosing to week 20
Immunogenicity | From dosing to week 20
  Number of anti-ALD1910 antibodies (ADA) and characterization of anti-ALD1910 ADA positive responses for neutralizing activity

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Australia